CLINICAL TRIAL: NCT06887517
Title: Chinese Rheumatism Biobank(CRB)
Status: Recruiting | Type: Observational
Sponsor: Chinese SLE Treatment And Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CSTAR010
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: systemic lupus erythematosus; major organ damage; progress of disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Antimalarials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood samples , from which DNA, RNA, serum, plasma, cfRNA, cfDNA, PBMC are isolated；
  2. Nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Antimalarial with or without oral glucocorticosteroid — Intervention one: Antimalarial and Oral Glucocorticosteroid, Prednisone or equivalent dose of glucocorticoid tapering: 0.5~0.6mg/kg/d(week 0~2), 0.3~0.4mg/kg/d(week 3~4), 15 mg/d(week 5~6), 10 mg/d(week 7~8), 7.5 mg /d(week 9~10), 5 mg/d(week 11~12), 2.5 mg/d(week 13~24), <2.5 mg/d(after week 24)；Hydroxychloroquin 6.5mg/kg/d but no more than 400mg/d for initial therapy, and reduce to 4~5mg/kg/d for maintenance therapy
  Intervention two: Antimalarial only. Hydroxychloroquin 6.5mg/kg/d but no more than 400mg/d for initial therapy, and reduce to 4~5mg/kg/d for maintenance therapy

SUMMARY:
Early prediction of major organ damage in SLE needs to dynamically track the evolution of SLE patients before and after the onset of major organ damage, and analyze the microscopic molecular evolution patterns synchronized with the macroscopic pathophysiological changes.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a complex autoimmune disease characterized by the presence of multiple autoantibodies in the serum and multisystemic damage.The clinical manifestations of SLE are highly heterogeneous, and damage to different organs appears gradually over time. Lupus nephritis (LN) and thrombocytopenia (TP) represent the most common major organ damage in SLE, with an incidence of about 30-40%; pulmonary arterial hypertension (PAH) is a rare but difficult complication of SLE. Pulmonary arterial hypertension (PAH) is a rare but intractable complication of SLE, which clinically manifests itself as a progressively worsening increase in pulmonary arterial pressure, and ultimately causes right heart failure or even death. Once combined with LN, TP, PAH and other important organ damage, the long-term prognosis and quality of life of SLE patients are severely impaired.

Some predictive models for the occurrence of organ involvement in SLE have been reported in previous studies. Among them, several incidence prediction models for lupus nephritis (LN) included demographic, clinical and laboratory indicators such as male, anti-dsDNA antibody positivity, age and duration of SLE onset, erythrocyte sedimentation rate, mucosal ulceration, proteinuria, hematuria, etc., with the area under the curve (AUC) of the prediction model of 0.707. A prediction model for incidence prediction of neuropsychiatric lupus (NPSLE) incorporated both patient disease and environmental indicators, including anti-dsDNA antibody positivity, anti-SSA antibody positivity, lymphocyte count, erythrocyte pressure volume, erythrocyte sedimentation rate, prealbumin, retinol-binding protein, creatine kinase isoenzyme MB, brain natriuretic peptide precursor, creatinine, indirect bilirubin, fibrinogen, ultrasensitive C-reactive protein, CO, and mild contamination, which had an AUC in the discovery and validation cohorts of up to 0.849-0.895. Our center team has developed 2 predictive models for the onset of SLE organ involvement: the SLE-associated pulmonary arterial hypertension (PAH) onset prediction model contains 5 clinical variables (acute/subacute cutaneous lupus, arthritis, renal involvement, thrombocytopenia, and interstitial lung disease) and 3 autoantibodies (anti-RNP antibody positivity, anti-Ro/SSA antibody positivity, and anti-La/SSB antibody positivity). La/SSB antibody positive). The above predictive models for the occurrence of SLE organ involvement basically used easily accessible clinical data, such as clinical manifestations and laboratory indicators, and the models were practical; however, most of the models were not constructed based on prospective cohorts, and some of the models were not validated in large-scale patient populations, so the predictive efficacy of the models is still unsatisfactory, and their clinical application is still difficult.

There is still a lack of effective biomarkers and prediction models for important organ damage in SLE. The fundamental problem is that there is no high-quality cohort of SLE patients before and after the onset of organ damage. Therefore, early prediction of vital organ damage in SLE can only be achieved by dynamically tracking the evolution of SLE patients before and after the onset of vital organ damage, and analyzing the microscopic molecular evolution patterns synchronized with the macroscopic pathophysiological changes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the 2012 SLICC classification criteria or 2019 ACR/EULAR classification criteria of SLE.
2. Disease Duration ≤2 years since SLE diagnosis at baseline
3. Non-Organ-Threatening Disease, including BILAG-2004 categories A/B/C in neurological, cardiopulmonary, gastrointestinal, ophthalmic, renal, or hematological domains

   Specifically excluded:

   Renal: Cellular casts, hematuria (>5 RBC/hpf), proteinuria (>0.5g/24hr), pyuria (>5 WBC/hpf), or biopsy-proven lupus nephritis Neuropsychiatric: Seizures, psychosis, organic brain syndrome, cerebrovascular events Cardiopulmonary: Pulmonary arterial hypertension, myocarditis, pulmonary hemorrhage Vasculitis: Ulcerative/necrotizing lesions or biopsy-proven vasculitis Hematologic: Hemolytic anemia, thrombocytopenia (<100×10⁹/L) No acute thromboembolic events within 3 months
4. Treatment History:

   No systemic corticosteroids, plasmapheresis, or IVIG within 3 months No biologics (e.g. belimumab, TNF-α inhibitors) within 3 months No cyclophosphamide or CD20 inhibitors within 6 months
5. Disease Activity: Clinical SLEDAI-2K >0 at screening/baseline

Exclusion Criteria:

1. SLE with coexisting other autoimmune or autoinflammatory diseases, including but not limited to rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, or psoriasis.
2. SLE with concurrent conditions requiring glucocorticoid therapy, such as asthma or Crohn's disease.
3. Pregnancy, planned pregnancy, or lactation.
4. SLE with major organ dysfunction at baseline , including: impaired consciousness or cognitive decline, renal insufficiency, cardiac insufficiency (NYHA Class 3 or 4), pulmonary hypertension or interstitial lung disease, uncontrolled infections
5. Inability to ensure compliance with long-term follow-up
6. Any condition deemed by investigators to compromise trial completion or pose significant risks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with systemic lupus erythematosus (SLE) at Peking Union Medical College Hospital, who met the inclusion/exclusion criteria and voluntarily provided written informed consent.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2033-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major organ involvement in SLE | From enrollment to the end of 60 months
  Occurrence of lupus nephritis, immune thrombocytopenia or pulmonary arterial hypertension.

SECONDARY OUTCOMES:
Occurrence of disease activity within 24 weeks | From enrollment to the end of 24 weeks
  Disease activity was defined as the presence of fever, alopecia, rash, arthritis, mucosal ulcers, myositis, pleurisy, pericarditis, decreased complement levels, or increased anti-ds-DNA antibody levels, etc.
Failure to meet DORIS remission criteria at the end of 24 weeks | From enrollment to the end of 24 weeks.
  DORIS stands for Definitions of remission in systemic lupus erythematosus. Clinical remission was defined as:
  1. cSLEDAI (SLEDAI-2K Clinical Indicator) = 0 (except for low complement and anti-dsDNA positivity)
  2. PGA <0.5 points
  3. No oral glucocorticoids
  4. Immunosuppressants (except CTX) and biologics are stable, antimalarials are available

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology and Clinical Immunology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing, Beijing Municipality, China